CLINICAL TRIAL: NCT02078102
Title: A Phase II Trial of Prostaglandin E2 Inhibition, Using Meloxicam, Plus Filgrastim for Mobilization of Autologous Peripheral Blood Stem Cells in Patients With Multiple Myeloma and Non-Hodgkin's Lymphoma
Brief Title: A Phase II Trial Using Meloxicam Plus Filgrastim in Patients With Multiple Myeloma and Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sherif S. Farag (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sherif S. Farag, Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0419; CA182947 (Other Grant/Funding Number: NCI); 1312925163 (Other: Indiana University IRB)
Record Dates: First submitted 2014-02-20; First posted 2014-03-05 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Meloxicam; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Meloxicam and Filgrastim will be administered in fixed doses to each patient enrolled on this study. The treatments will be administered in a staggered dose schedule for a total treatment duration of 7 days prior to apheresis.
  15 mg tablets of Meloxicam will be taken orally for 5 consecutive days.
  10 µg/kg of Filgrastim will be subcutaneously injected for 5 consecutive days. Filgrastim may be subcutaneously injected for an additional 3 days if patients do not meet the primary endpoint for cell collection.
  Interventions: Drug: Meloxicam; Drug: Filgrastim

INTERVENTIONS:
Drug: Meloxicam — 15 mg tablets of Meloxicam will be taken orally in the morning, with or without food.
  Other Names: Mobic
Drug: Filgrastim — Filgrastim will be subcutaneously injected in one or two sites at home.
  Other Names: Neupogen

SUMMARY:
The trial is an open label Simon optimal two-stage Phase II trial of fixed doses of oral meloxicam and subcutaneous filgrastim to assess the safety and efficacy in mobilizing autologous peripheral blood stem cells (PBSC) from multiple myeloma (MM) and non-Hodgkin's lymphoma (NHL) patients planning to undergo high-dose chemotherapy with stem cell support. Clinical data regarding the cellular composition and function of the graft mobilized by this combination will be obtained.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study:

1. Has provided written informed consent prior to completing any study procedures.
2. Patients must have a previously documented histologic diagnosis of multiple myeloma (MM) or non-Hodgkin's lymphoma (NHL), and be eligible to undergo autologous PBSC transplantation on institutional protocols.

   1. Multiple myeloma should be in first or second partial response or better, as defined by International Myeloma Working Group criteria.50
   2. Non-Hodgkin's lymphoma must be in either first or second partial response or better and have any one of the following histologies:

      * Diffuse large B cell lymphoma
      * Transformed lymphoma
      * Mantle cell lymphoma
      * Follicular lymphoma (any grade)
      * Peripheral T cell lymphoma
3. Age ≥18 to ≤75 years at time of consent.
4. Karnofsky performance status of at least 70%.
5. Adequate organ function defined as:

   1. Left ventricular ejection fraction ≥45%
   2. Corrected DLCO ≥50%
   3. Serum bilirubin, AST (aspartate aminotransferase) and ALT(alanine aminotransferase) ≤ twice the upper limit of normal
   4. Serum creatinine ≤ 2.0 mg/dl
   5. Urine M-protein ≤1 g/24 hours (MM patients only)
6. No prior attempt at mobilizing PBSC.
7. Patients must be at least 4 weeks from last cytotoxic chemotherapy (including alkylating, anthracyclines, epipodophylatoxins, and platinum drugs), or immunomodulatory drugs (including lenalidomide or pomalidomide, or related derivatives) at time of treatment on this protocol.
8. Patients must be at least 2 weeks from last treatment with a proteasome inhibitor (e.g., bortezomib, carfilzomib) at time of treatment on this protocol.
9. Patients must be negative for HIV.
10. Women of childbearing potential must have a negative pregnancy test (urine or serum) and must not be lactating at the time of informed consent.

    1. Women and men must use adequate birth control while taking part in this study (such as a condom or diaphragm with contraceptive cream/jelly, birth control pills, Norplant, abstinence (no sexual intercourse) or surgical sterilization.

Exclusion Criteria:

Exclude a patient if any of the following conditions are observed:

1. Patients must not have received radiation therapy within the past 4 weeks, and not to more than 20% of hematopoiesis forming bones (spine, pelvis and proximal long bones).
2. Patients must not have active central nervous system involvement.
3. Patients must not have a prior autologous, syngeneic or allogeneic hematopoietic stem cell transplant.
4. Patients must not have received prior bone seeking radionuclides.
5. Patients must not have received myeloid growth factors within 2 weeks before mobilization attempt on this study.
6. Patients must not have taken nonsteroidal antiinflammatory drugs (NSAID) in the past 14 days before treatment on this protocol.
7. Patients must not have nor had active or recent peptic ulcer disease within the past 6 months.

   a) Patients with active significant symptoms of dyspepsia will be excluded.
8. Patients with a history of asthma will be excluded because of the potential for NSAID to precipitate asthma in these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, M.D., Ph.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Patterson AM, Zhang S, Liu L, Li H, Singh P, Liu Y, Farag SS, Pelus LM. Meloxicam with Filgrastim may Reduce Oxidative Stress in Hematopoietic Progenitor Cells during Mobilization of Autologous Peripheral Blood Stem Cells in Patients with Multiple Myeloma. Stem Cell Rev Rep. 2021 Dec;17(6):2124-2138. doi: 10.1007/s12015-021-10259-y. Epub 2021 Sep 12. PMID 34510361

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Myeloma: This is for the patients with Multiple Myeloma.
  Meloxicam and Filgrastim will be administered in fixed doses to each patient enrolled on this study. The treatments will be administered in a staggered dose schedule for a total treatment duration of 7 days prior to apheresis.
  15 mg tablets of Meloxicam will be taken orally for 5 consecutive days.
  10 µg/kg of Filgrastim will be subcutaneously injected for 5 consecutive days. Filgrastim may be subcutaneously injected for an additional 3 days if patients do not meet the primary endpoint for cell collection.
  Meloxicam: 15 mg tablets of Meloxicam will be taken orally in the morning, with or without food.
  Filgrastim: Filgrastim will be subcutaneously injected in one or two sites at home.
- Non Hodgkins Lymphoma: This is for the patients with Non Hodgkins Lymphoma.
  Meloxicam and Filgrastim will be administered in fixed doses to each patient enrolled on this study. The treatments will be administered in a staggered dose schedule for a total treatment duration of 7 days prior to apheresis.
  15 mg tablets of Meloxicam will be taken orally for 5 consecutive days.
  10 µg/kg of Filgrastim will be subcutaneously injected for 5 consecutive days. Filgrastim may be subcutaneously injected for an additional 3 days if patients do not meet the primary endpoint for cell collection.
  Meloxicam: 15 mg tablets of Meloxicam will be taken orally in the morning, with or without food.
  Filgrastim: Filgrastim will be subcutaneously injected in one or two sites at home.
Period: Overall Study
Arm/Group | Multiple Myeloma | Non Hodgkins Lymphoma
Started | 25 | 13
Completed | 23 | 12
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple Myeloma | Non Hodgkins Lymphoma | Total
Number analyzed (Participants) | 25 | 13 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 11 | 27
  >=65 years | 9 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (8.6) | 51.2 (16.1) | 57.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 11 | 33
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 21 | 10 | 31
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Disease Status at Registration [Count of Participants; unit: Participants] — Multiple Myeloma response was determined by the International Myeloma Working Group criteria (based on serum, urine and blood markers) and the Non-Hodgkin's response was determine by the Lymphoma Response Criteria (based on metabolic and radiographic criteria). Entry criteria for the study required a partial response or better for entry into the study.
  Participants
    Partial Response | 19 | 0 | 19
    Partial Response without prior Complete Response | 0 | 1 | 1
    Very Good Partial Response | 5 | 1 | 6
    Complete Remission | 1 | 9 | 10
    Complete Remission Confirmed | 0 | 1 | 1
    Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Mobilize and Collect at Least Half of the Total Target CD34+ Cell Dose in the First Apheresis
Description: Percent of patients who mobilize and collect at least half of the total target CD34+ cell dose in the first apheresis with binomial exact confidence intervals according to disease:
  Multiple myeloma patients: percent of patients with >= 5x106 CD34 cells/kg in the first day's apheresis. Non-Hodgkin's lymphoma patients: percent of patients with >= 2.5x106 CD34 cells/kg in the first day's apheresis.
Time Frame: within 100 days of transplant
Population: Patients with available post-transplant CD34+ results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Multiple Myeloma | Non Hodgkins Lymphoma
Number analyzed (Participants) | 25 | 12
percentage of participants | 32.0 [15.0 to 53.5] | 58.3 [27.7 to 84.8]

2. Secondary Outcome: Number of Patients With Treatment Related Adverse Events Grade 3 or Higher for Nonhematological Toxicity
Description: Number of unique patients who had a treatment related (possible, probable or definite) non-hematological adverse event that was graded 3 or greater using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: within 100 days of transplant
Population: All patients who received a transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma | Non Hodgkins Lymphoma
Number analyzed (Participants) | 25 | 13
Participants | 0 | 0

3. Secondary Outcome: Summary Statistics for Graft Composition of Peripheral Blood Stem Cell Collection at Each Time Point
Description: Mean and Standard Deviation of the Graft Composition of Peripheral Blood Stem Cell Collection (CD34 (x10^6cells/kg)) at each time point collected during Cycle 2.
Time Frame: Cycle 2, Days 1-4, within 100 days of transplant
Population: Patients with available post-transplant CD34 (x10^6/kg) data.
Measure: Mean (Standard Deviation); unit: x10^6cells/kg
Arm/Group | Multiple Myeloma | Non Hodgkins Lymphoma
Number analyzed (Participants) | 25 | 12
x10^6cells/kg
  Cycle 2 Day 1 | 3.42 (2.72) | 3.22 (2.20)
  Cycle 2 Day 2: number analyzed (Participants) | 23 | 9
  Cycle 2 Day 2 | 4.92 (2.86) | 3.51 (2.67)
  Cycle 2 Day 3: number analyzed (Participants) | 9 | 3
  Cycle 2 Day 3 | 2.63 (1.70) | 0.89 (0.45)
  Cycle 2 Day 4: number analyzed (Participants) | 2 | 1
  Cycle 2 Day 4 | 1.55 (0.35) | 0.90 (NA) — Only 1 patient had a result at this time point and the standard deviation was not calculated.

4. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. The median and 95% confidence intervals will be provided. Only patients with neutrophil engraftment will be included.
Time Frame: within 100 days of transplant
Population: All patients who had a transplant and engrafted. All patients were analyzed together since the definition for neutrophil engraftment is the same regardless of disease and only the time until overall neutrophil engraftment was the outcome of interest.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Treatment Group: Meloxicam and Filgrastim will be administered in fixed doses to each patient enrolled on this study. The treatments will be administered in a staggered dose schedule for a total treatment duration of 7 days prior to apheresis.
  15 mg tablets of Meloxicam will be taken orally for 5 consecutive days.
  10 µg/kg of Filgrastim will be subcutaneously injected for 5 consecutive days. Filgrastim may be subcutaneously injected for an additional 3 days if patients do not meet the primary endpoint for cell collection.
  Meloxicam: 15 mg tablets of Meloxicam will be taken orally in the morning, with or without food.
  Filgrastim: Filgrastim will be subcutaneously injected in one or two sites at home.
Arm/Group | Treatment Group
Number analyzed (Participants) | 34
days | 13.0 [12.0 to 14.0]

5. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive Complete Blood Counts (CBCs) obtained on different days after transplantation during which the platelet count is at least 20 x109/l. The CBCs obtained should be at least seven days after the most recent platelet transfusion. The median and 95% confidence intervals will be provided. Only patients achieving platelet engraftment will be included.
Time Frame: within 100 days of transplant
Population: All patients who received a transplant and engrafted. All patients were analyzed together since the definition for platelet engraftment is the same regardless of disease and only the time until overall platelet engraftment was the outcome of interest.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment Group
Number analyzed (Participants) | 34
days | 16.5 [13.0 to 19.0]

ADVERSE EVENTS:
Time Frame: up to 100 days post-transplant
Arm/Group | Multiple Myeloma | Non Hodgkins Lymphoma
All-Cause Mortality (participants affected / at risk) | 4/25 | 1/13
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/13
Other Adverse Events (participants affected / at risk) | 10/25 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multiple Myeloma (N=25) | Non Hodgkins Lymphoma (N=13)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Multiple Myeloma (N=25) | Non Hodgkins Lymphoma (N=13)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 6
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Pain (General disorders) | 1 | 2
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT02078102/Prot_SAP_000.pdf